CLINICAL TRIAL: NCT04659265
Title: The Effect of a Wrong Suspected Diagnosis of a Pre-treating Physician on the Correctness of the Final Diagnosis
Brief Title: A Priori Diagnosis and Diagnostic Errors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Stephan Marsch, Professor of Intensive Care, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4031-Sim-1
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Error Disclosure; Diagnoses Disease; Simulation of Physical Illness
Keywords: diagnostic error; presumptive diagnosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants not aware of the study goal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No suspected diagnosis (control group) (Active Comparator): Participants receive the information that the pre-treating physician thought that the patient is suffering from a medical emergency (no diagnosis).
  Interventions: Other: Suspected diagnosis of a pre-treating physician
- Correct suspected diagnosis (Active Comparator): Participants receive the information that the pre-treating physician thought that the patient is suffering from an acute myocardial infarction (correct diagnosis).
  Interventions: Other: Suspected diagnosis of a pre-treating physician
- Wrong suspected diagnosis (Active Comparator): Participants receive the information that the pre-treating physician thought that the patient is suffering from a pulmonary embolism (wrong diagnosis).
  Interventions: Other: Suspected diagnosis of a pre-treating physician

INTERVENTIONS:
Other: Suspected diagnosis of a pre-treating physician — Participants receive the information that the pre-treating physician thought the patient is suffering from a medical emergency (no diagnosis), an acute myocardial infarction (correct diagnosis) or a pulmonary embolism (wrong diagnosis)

SUMMARY:
This is a prospective randomized single-blind simulator-based trial. 156 4th year medical students were randomised to receive one of three different suspected diagnoses of a pre-treating physician (no diagnosis, myocardial infarction, pulmonary embolism) prior to the task to make a focussed assessment and perform first management steps in a patient presenting to the emergency department. The patient (simulator) suffered from an acute myocardial infarction. Video recordings were obtained during simulation and used for data analysis. Primary endpoint was the participants' final presuptive diagnosis.

DETAILED DESCRIPTION:
Methods:

Study design:

This is a prospective randomized controlled single-blind trial, the participants not being aware of the purpose of the study. The trial was approved by the regional ethical committee (EKNZ 85/04) and all participants gave written informed consent.

Participants:

Medical students in their 4th year at the University of Basel, Switzerland were offered to participate in voluntary workshops at the simulator centre of the medical intensive care unit of university of Basel hospital. The present study was conducted as part of these workshops.

At the beginning of the workshop participants were asked to fill in a questionnaire. The questionnaire included a) the Big Five personality traits (neuroticism, extraversion, openness, agreeableness, conscientiousness) (McCrae 1992); b) Rosenberg's self-esteem scale(Colani); c) the task to diagnose the cardiac rhythm in 12 one-lead ECG rhythms strips (each correct diagnosis was counted as one point resulting in a maximum of 12 attainable points); d) the task to list the typical symptoms of an acute myocardial infarction in bullet point form (each of the following items were counted as one point resulting in a maximum of 6 attainable points: chest pain; radiation of the pain; pain described as constricting, compressing, or squeezing; at least one accompanied vegetative symptom; dyspnoea; and fear); and e) the task to list the typical signs symptoms of 4 further medical emergencies (anaphylactic shock, trauma management, cardiac arrest, syncope) in bullet point form (answers were coded using a predefined checklist).

Simulator and Scenario:

The study was conducted using a patient simulator. All participants received a standardised instruction of the patient simulator (human patient simulator, Leardal SimMan®). This simulator's features include among others palpable pulses, spontaneous breathing with visible thoracic excursions, spontaneous movements of the eye lids and a speaker in the mannequin's head that broadcasts the voice of a remote operator, allowing for verbal interaction with the participants. For the present trial, the operator was an experienced physician.

For the study scenario participants were given the role of a resident-on-call in the emergency department and were instructed by a senior physician (confederate) to triage a newly arrived patient. Upon entering the simulator room, the participants encountered the patient (simulator) lying on a bed and dressed in a hospital gown. Participants were assisted by a confederate nurse. The nurse was instructed to display a helpful manner, to act only on command, but not to interfere in any way with the assessment and history taking.

Intervention:

All participants performed the scenario on their own and faced a patient with a simulated acute myocardial infarction. Participants were randomized (computer-generated numbers) to three versions of the scenario. The three versions differed only in the reply of the patient to the initial question about the reason for his visit. The patient volunteered that he had phoned his family physician because of acute chest pain and dyspnoea. The family physician had recommended urgent visit of the emergency department because he judged the situation as 1) medical emergency (control group with no à priori diagnosis); 2) acute myocardial infarction (correct à priori diagnosis group); or, 3) acute pulmonary embolism (wrong à priori diagnosis group). Apart from this randomly allocated initial information, the scenario was identical in all groups: until the end of the scenario, the patient only spoke when asked a question and all answers were given according a pre-scripted answer check-list (table) Participants of the groups with no à priori diagnosis and correct à priori diagnosis were given 4 minutes study time. Participants of the group with wrong diagnosis were given one additional minute (i.e. 5 minutes study time) to compensate for probing the given diagnosis. At the end of the study time, the senior physician entered the room and announced that he required the participant to temporarily leave his/her patient to help with another emergent case. The participants were then asked on their presumptive diagnosis and which measures, if any, the nurse should take during their temporary absence during the next couple of minutes.

Data analysis:

Data analysis was performed using video recordings obtained during simulations. Video recordings were analysed independently by two trained raters who noted all questions asked and all measures taken by the participant. Inter-observer differences were solved by jointly re-watching the video recordings.

Statistics:

The primary endpoint was a correct presumptive diagnosis of an acute myocardial infarction or acute coronary syndrome when asked at the end of the scenario by the senior physician or when previously revealed to the patient and/or the nurse. Mentioning the correct diagnosis as possible differential diagnosis was rated as correct diagnosis. A co-primary endpoint was the composite endpoint of a correct presumptive diagnosis OR ordering a 12-lead ECG, the rationale being that a timely 12-lead ECG will most likely prevent harm to a patient not correctly triaged as suffering from acute myocardial infarction.

Secondary endpoints were the number and kind of questions asked during history taking; probing of the à priori diagnosis; measures taken during assessment; and the results of the questionnaire. Results of the knowledge part of the questionnaire are reported as percentages of the attainable maximum.

A 20% difference in the primary outcome was considered to be of medical relevance- A power analysis revealed that approximately 150 teams (50 per group) had to be included to detect this difference with a power of 0.9 at the 0.05 significance level.

Statistical analysis was performed by SPSS (version 25). Non-parametric ANOVA, Mann-Whitney test, chi-square test, Univariate and Multivariate regression analysis, and Cohen's kappa were used as appropriate. A p < 0.05 was considered to represent statistical significance. Data are reported as median [Interquartile range {IQR}] unless otherwise stated.

ELIGIBILITY:
Inclusion Criteria:

* 4th year medical students and physicians taking part in simulation workshops

Exclusion Criteria:

* no consent given to video-tape simulation and analyse vide recordings for scientific purpose

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Correct diagnosis | 5 minutes
  Correct presumptive diagnosis

SECONDARY OUTCOMES:
number and kind of questions asked during history taking | 5 minutes
  number and kind of questions asked during history taking
probing of the à priori diagnosis | 5 minutes
  questions related to the given à priori diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Marsch, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Department of Medical Intensive Care; University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No
The core data of the study are video-recordings of a simulation. These data cannot be shared as they are strictly confidential as indicated in the participants' consent forms.